CLINICAL TRIAL: NCT04272138
Title: Feasibility of Using a Mobile App (i.e., Calm) to Decrease Overall Stress in Middle-aged (i.e., 40-64 Years) Men and Women Who Report High Stress (>15 on PSS)
Brief Title: A Brief App-based Mobile Health and Well-being Intervention Among Middle-aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00011219
Record Dates: First submitted 2020-01-13; First posted 2020-02-17 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Meditation; Control Group

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm Meditation (Experimental): Participants in the intervention group will be exposed to 10 minutes per day of meditation via a smartphone application for 4 weeks. Participants will log their meditation participation in an online weekly log.
  Interventions: Behavioral: Calm Meditation
- Educational Podcast Control (Active Comparator): Participants in the control group will be exposed to 10 minutes per day of health education podcasts via a smartphone application for 4 weeks. Participants will log their podcast participation in an online weekly log.
  Interventions: Behavioral: Educational Podcast Control

INTERVENTIONS:
Behavioral: Calm Meditation — The intervention will run for 4-weeks. Participants will complete the 30 day, "How to Meditate" meditation series that provides daily 10-minute meditations. Throughout the intervention, participants will be sent reminder emails via REDCap to participate in their assigned practice sessions participants and will complete online weekly participation logs via REDCap. Additionally, they will answer one, multiple-choice ecological momentary assessment question, randomly, 3x per day via test message assessing how one currently feels. Participants will complete baseline and post-intervention measures of the Perceived Stress Scale, Hospital Anxiety and Depression Scale, Mindfulness Attention Awareness Scale, International Physical Activity Questionnaire, Salzberg Stress Eating Scale, Brief Cope, and Brief Resilience Scale. Following these measures, participants will be asked to complete a satisfaction questionnaire (week 5) and have the opportunity to volunteer for a short phone interview.
  Arms: Calm Meditation
Behavioral: Educational Podcast Control — The intervention will run for 4-weeks. Control group participants will listen to daily 10-minute health education podcasts. Throughout the intervention, participants will be sent reminder emails via REDCap to participate in their assigned practice sessions and participants will complete online weekly participation logs via REDCap. Additionally, they will answer one, multiple-choice EMA (ecological momentary assessment) question, randomly, 3x per day via test message assessing how one currently feels. Participants will complete baseline and post-intervention measures of the Perceived Stress Scale, Hospital Anxiety and Depression Scale, Mindfulness Attention Awareness Scale, International Physical Activity Questionnaire, Salzberg Stress Eating Scale, Brief Cope, and Brief Resilience Scale. Following these measures, participants will be asked to complete a satisfaction questionnaire (week 5) and have the opportunity to volunteer for a short phone interview.
  Arms: Educational Podcast Control

SUMMARY:
The purpose of this study is to determine the preliminary effects of using a mobile app (i.e., Calm) to decrease overall stress in middle-aged (i.e., 40-64 years) men and women who report high stress (greater than 15 on PSS).

The study design is a randomized control trial with baseline, post-intervention (4 weeks from baseline), and follow-up phone interview (5 weeks from baseline) assessments. Middle-aged adults will be randomized to either a Calm meditation Intervention group or an attention control podcast group. Participants will be randomized after the completion of baseline and informed consent.

Specific aim 1: Determine the feasibility (acceptability, demand) of using CALM app at least 10 min/day to reduce stress (greater than 15 on Perceived Stress Scale [PSS]) in middle-aged men and women.

Benchmarks for feasibility: (acceptability) Recruitment greater than 40 percent men; greater than 75 percent satisfied with intervention; 75 percent perceive daily meditation and app components as appropriate and useful; (demand) Retention of men greater than 75 percent; greater than 80 percent adherence (minutes/week) to the meditation intervention.

Specific aim 2: Explore the preliminary effect of meditation using Calm on overall perceived stress as compared to the health education group.

Specific aim 3: Explore the preliminary effect of meditation using Calm on anxiety and depression.

Specific aim 4: Explore gender as a moderator of the effect of meditation using Calm on stress.

Specific aim 5: Explore the mediators of mindfulness, physical activity, eating, and coping behaviors on stress, anxiety and depression using Calm for meditation.

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited during winter/spring 2020. Interested participants will be directed to a REDCap link to complete an online eligibility screener. The screener will take approximately 10 minutes to complete (See Eligibility Survey). The survey will be free, voluntary, and available online. Participants will be allowed to skip questions in the survey.

Eligibility: Once eligibility is determined; participants will be sent an informed consent and baseline questionnaire via a REDCap link. This measure should take approximately 25 minutes to complete (See Informed Consent and Baseline Questionnaires). Once Informed Consent is signed and the Baseline Questionnaires are complete, participants will be randomized via an online randomizer (i.e., randomizer.com) to either an attention control podcast group or the Calm meditation group. Ineligible participants will be sent an email notifying their status and why.

Enrollment: The Research Team will email the intervention participants that will include instructions to download Calm (See Participant Scripts). The control participants will be emailed instructions to download the podcast app (See Participant Scripts).

Intervention: The intervention will run for 4-weeks. Intervention participants will complete the 30 day, "How to Meditate" meditation series that provides daily 10-minute meditations and the control group will listen to daily 10-minute health education podcasts. Throughout the intervention, both groups will be sent reminder emails via REDCap to participate in their assigned practice sessions (see Participant Scripts) participants will complete online weekly participation logs via REDCap. Additionally, they will answer one, multiple choice EMA (ecological momentary assessment) question, randomly, 3x per day (between 8am and 8pm) via test message assessing how one currently feels (see Study Questionnaires).

Tracking: Participation in the Calm meditations will be tracked (meditation name, time of day, and time spent in meditation) by weekly REDCap participation logs and the Calm team.

Post-intervention: Post-intervention questionnaires and the satisfaction survey will be emailed to intervention and control participants via a link from REDCap (See Post-intervention questionnaires). The post-intervention survey will take about 25 minutes and the satisfaction survey will take about 10 minutes.

Post-intervention interview: Post-intervention phone interviews will be conducted the week following the end of the intervention (week 5) to no more than 20 participants in each group and take about 15-20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Age 40-64
* Able to read/understand English
* Have access to a smartphone on a daily basis
* A score of 15 or higher on the Perceived Stress Scale (PSS)
* Willing to be randomized
* Willing to download a mobile application

Exclusion Criteria:

* Have consistently practiced mindfulness meditation within the last 12 months
* Currently using the Calm app or another meditation app
* Currently prescribed mental health or mood medication
* Low levels of stress (i.e., less than a score of 15 assessed with the Perceived Stress Scale)
* Currently reside outside the United States

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Feasibility: Acceptability | Measured 1x at post-intervention about experience in study, about 4 weeks.
  Acceptability will be measured using a satisfaction survey at the end of the study, following all other measures (satisfied with the intervention and perceive daily meditation and app components as appropriate and useful)
Feasibility: Demand | 1x at post-intervention about participation time in study (4 weeks total)
  Demand will be measured using the subjective usage data (weekly participation logs measuring adherence (minutes/week) and the objective app usage data (data collected by the app measuring adherence (minutes/week) to the meditation intervention).

SECONDARY OUTCOMES:
Stress | Change from baseline (week 0) to post-intervention (week 4)
  Stress will be measured using the Perceived Stress Scale -10 item, with scores ranging from 10-40) and a higher score indicates a worse outcome.
Anxiety | Change from baseline (week 0) to post-intervention (week 4)
  Anxiety will be measured using the Hospital Anxiety and Depression Scale, with scores ranging from 0-21, and a higher score indicates a worse outcome.
Depression | Change from baseline (week 0) to post-intervention (week 4)
  Depression will be measured using the Hospital Anxiety and Depression Scale, with scores ranging from 0-21, and a higher score indicates a worse outcome.
Gender as moderator of stress | Change from baseline (week 0) to post-intervention (week 4)
  Self-reported gender
Mindfulness as a mediator of stress | Change from baseline (week 0) to post-intervention (week 4)
  Mindfulness will be measured using the Mindful Attention Awareness Scale, with scores ranging from 15-90, and a higher score indicates a better outcome.
Physical Activity as a mediator on stress, anxiety, and depression | Change from baseline (week 0) to post-intervention (week 4)
  Physical activity will be measured using the International Physical Activity Questionnaire, when a higher score indicates a better outcome.
Eating as a mediator on stress, anxiety, and depression | Change from baseline (week 0) to post-intervention (week 4)
  Eating will be measured using the Salzburg Stress Eating Scale, with scores ranging from 5-100, and a higher score indicates a worse outcome.
Coping behaviors as a mediator on stress, anxiety, and depression | Change from baseline (week 0) to post-intervention (week 4)
  Coping behaviors will be measured using the Brief COPE Inventory, with scores ranging from 2-8, and a higher score indicates a better outcome.
Resilience | Change from baseline (week 0) to post-intervention (week 4)
  Resilience will be measured using the Brief Resilience Scale, with scores ranging from 1-5, and a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huberty, PhD, Study Chair — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laird B, Puzia M, Larkey L, Ehlers D, Huberty J. A Mobile App for Stress Management in Middle-Aged Men and Women (Calm): Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 May 24;6(5):e30294. doi: 10.2196/30294. PMID 34989677